CLINICAL TRIAL: NCT05607511
Title: Improvement in Eczema and the Safety of Microbiome Baby Immunity Formula (SIM03) on Childhood Eczema Development - A Pilot Study
Brief Title: GB-EZ-SIM03 Probiotics Study for Childhood Eczema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ting-fan Leung, Alice Ho Miu Ling Nethersole Charity Foundation Professor of Paediatrics, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG2217044
Record Dates: First submitted 2022-10-28; First posted 2022-11-07 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Eczema
Keywords: Eczema; Probiotics; Open-label study; Microbiome; Children
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Intervention Model Description: Single-group, open-label interventional clinical trial
Masking Description: Masked laboratory staff about the clinical details and disease-related information of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active probiotics arm (Experimental): The SIM03 (supplied by GenieBiome Limited and produced under Good Manufacturing Practice, GMP) contains a blend of naturally occurring food-grade Bifidobacterium strains (1 billion CFU in 1 sachet). Recruited subjects will receive one sachet of baby immunity formula SIM03 twice daily for 3 months.
  Interventions: Other: Probiotics baby immunity formula (SIM03)

INTERVENTIONS:
Other: Probiotics baby immunity formula (SIM03) — Daily oral intake of a probiotics sachet

SUMMARY:
Eczema is the most prevalent chronic skin disease in young children, and skin infection is commonly seen during eczema flare. Dysbiosis is increasingly recognised in the stool and skin of these patients. It is a common practice for parents to start these eczematous children on probiotics, but there is limited evidence if this treatment works in young patients. This single-centre, open-label clinical trial aims to investigate the benefits of a 3-month treatment of young children with eczema with a new probiotics called microbiome baby immunity formula (SIM03). Study outcomes include eczema severity, quality of life, biophysical measures of the skin and gastrointestinal symptoms, while adverse events related to this probiotics treatment will be monitored. The effects of this intervention on stool microbiome will also be analysed.

DETAILED DESCRIPTION:
Eczema is a common chronic skin disease that affects a substantial part of population. The associated economic burden was estimated to cost more than $5 billion per year with the rising prevalence of this disease worldwide. A 2016 nation-wide study in China reported that 12.9% of children (1-7 years) were diagnosed with eczema. Growing evidence has shown that atopic dermatitis and/or eczema would increase the risk of several diseases' development, including stroke, myocardial infarction, unstable angina, atrial fibrillation, and cardiovascular death.

Except variation of clinical symptoms including dryness and itchy skin in eczema patients, gastrointestinal symptoms were also reported by children with atopic eczema, such as abdominal pain, abdominal distension, diarrhoea, constipation, vomiting and regurgitation. Unique gastrointestinal microflora pattern has also been observed in atopic dermatitis/ eczema patients when compared with healthy controls: decreased Bifidobacterium and Enterococci, especially Bifidobacterium bifidum and Bifidobacterium longum, and increased Faecalibacterium have been observed. Therefore, gastrointestinal microflora can serve as the disease indicator of eczema.

The development of gut microbiota starts before birth. The infant's microbiome can impact on human health in later life. To prevent disease, we need to nip it in the bud. Emerging evidence suggests that gut microbiota modulation can largely affect host immune functions in children and adults.

To date, no baby formula is specific for alleviating eczema-related symptoms for small children. GenieBiome Limited, a microbiome research-based company in Hong Kong developed a unique oral microbiome formula (baby immunity formula, SIM03) to prevent or treat gut dysbiosis and eczema development. SIM03 contains a blend of naturally occurring two food-grade probiotics strains, two prebiotics and two postbiotics. The two probiotics belong to food-grade Bifidobacterium, which is an important group of probiotic cultures commonly used in food products. Especially, research showed that Bifidobacterium could displace the proteolytic bacteria causing diarrhoea and recommended the administration of bifidobacteria to infants suffering from this symptom. Whereas the two prebiotics belong to food-grade oligosaccharides, which have been already used in food products. The two postbiotics belong to the acetates, which are also food grade and allowed to add in the foods.

We hypothesize that the gut microbiota of children with eczema can be modulated to decrease the severity of eczema related symptoms and the condition can be improved. A pilot study is proposed to assess the effect and safety of SIM03 on eczema severity, gut microbiome and GI symptoms of the children with eczema.

HYPOTHESIS We hypothesize that the microbiome baby immunity formula (SIM03) will lead to the improvement of eczema symptoms in children 1-5 years of age.

OBJECTIVES

1. To examine the effects of SIM03 in modulating gut microbiota, and improving the eczema severity, stool frequency/consistency in children aged 1-5 years old who have eczema;
2. To evaluate the safety of SIM03 by assessing the parent-reported adverse events in children aged 1-5 years old who have eczema in 1-5 years old children.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 1 to 5 years old with physician-diagnosed eczema according to Hanifin and Rakja criteria [22,23];
2. One of the parents or legal guardian (no mental illness or dementia, etc. that will hinder their ability to undertake informed consent) will provide written informed consent.

Exclusion Criteria:

1. Children with other documented chronic and clinically significant dermatologic diseases, such as erythra, that may interfere with evaluation of cutaneous microbiome. Common transient conditions such as acne are permissible.
2. Children with eczema who have taken antibiotics, probiotics or prebiotics in supplement, including but not limited to growing-up milk formula and infant's supplementary food within three months prior to inclusion.
3. Children with eczema who require systemic immunosuppressive treatments (e.g. corticosteroid, azathioprine, biologics) within six months prior to recruitment.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Total score for SCORing Atopic Dermatitis (SCORAD) | 3 months
  Combined endpoint
Stool frequency | 3 months
  Combined endpoint
Stool consistency | 3 months
  Combined endpoint

SECONDARY OUTCOMES:
Subjective SCORAD score | 3 months
  Disease severity
Objective SCORAD score | 3 months
  Disease severity
The change of stool frequency | 3 months
  Stool condition
The change of stool consistency assessed using Bristol Stool Chart | 3 months
  Stool condition
Quality of life assessment using a skin-specific Children's Dermatology Life Quality Index (CDLQI) and Infants' Dermatitis Quality of Life Index (IDQOL) | 3 months
  Quality of life related to eczema
Changes in faecal microbial profiling | 3 months
  Gut microbiome
The biophysical condition of skin as measured by TransEpidermal Water Loss | 3 months
  Skin biophysical parameters
The biophysical condition of skin as measured by Skin Hydration | 3 months
  Skin biophysical parameters
Adverse events reported during the study period | 3 months
  Monitoring of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Paediatrics, Prince of Wales Hospital, 30-32 Ngan Shing Street, Shatin, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
No need to disclose individual study data in this simple open-label clinical trial, thus it will report only the aggregate and summary of study findings from participants.